CLINICAL TRIAL: NCT05644158
Title: Effect of Different Treatment Strategies on Mitochondrial Function in Peripheral Arterial Disease - a Randomized Controlled Trial
Brief Title: Mitochondrial Function in Peripheral Arterial Disease
Acronym: MIVA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1194/2019
Record Dates: First submitted 2022-11-07; First posted 2022-12-09 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Peripheral Arterial Disease; Cardiovascular Diseases
Keywords: mitochondrial function; respirometry; near infrared spectroscopy; endothelial dysfunction; peripheral arterial disease; exercise training; revascularisation
MeSH Terms: conditions — Peripheral Arterial Disease; Cardiovascular Diseases | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled trial
  1. Exercise group
  2. Revascularization group
  3. Healthy control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise group (Active Comparator): Patients with intermittent claudication will receive conservative treatment with monitored exercise training for a total of 12 weeks (home-based training, minimum of three times a week, documented by using a diary with documentation of the type, the intensity and the duration of the training as well as by using a physical activity monitoring system (Move 4, Karlsruhe, Germany).
  Interventions: Other: Exercise therapy
- Revascularization group (Active Comparator): will receive revascularization of the underlying atherosclerosis lesion of the superficial femoral artery. Depending on the exact morphology of the lesion, patients with short superficial femoral artery lesions (<25 cm) will be subdivided into group 2A with endovascular treatment and patients with long superficial femoral artery lesions (>25 cm) will be subdivided into group 2B with open surgical treatment
  Interventions: Procedure: Revascularization
- Healthy control group (No Intervention): Patients undergoing surgery for symptomatic varicose veins with excluded PAD will serve as a control group.

INTERVENTIONS:
Procedure: Revascularization — Depending on the exact morphology of the lesion, patients with short superficial femoral artery lesions (<25 cm) will be subdivided into group 2A with endovascular treatment (percutaneous transluminal angioplasty with or without stenting) and patients with long superficial femoral artery lesions (>25 cm) will be subdivided into group 2B with open surgical treatment (femoropopliteal bypass) .
  Arms: Revascularization group
Other: Exercise therapy — Home-based monitored exercise training (walking), 3 times a week, monitored with log book and activity sensors.
  Arms: Exercise group

SUMMARY:
The aim of this study is to investigate the effect of different treatment strategies on mitochondrial function and to correlate in-vitro results to findings from in-vivo measurements of mitochondrial function. The authors hypothesize that interventional revascularization and therefore the restoration of blood and oxygen supply is more relevant to mitochondrial function compared to the effect of exercise training.

DETAILED DESCRIPTION:
Resulting from a chronic narrowing of arteries by atherosclerotic lesions, the leading clinical symptom of peripheral arterial disease (PAD), a walking induced pain, reduces quality of life of patients. Affected muscle regions are altered by a characterized myopathy and mitochondria are known to play a crucial role in this pathophysiological mechanism. There are different methodological approaches to investigate mitochondrial function in-vivo as well as in-vitro. Regarding our own preliminary data, mitochondria are known to recover after successful revascularization. The effect of different treatment strategies on mitochondrial function and the correlation of in-vitro to clinical more applicable in-vivo methods was understudied so far.

The overall aim of this study is to investigate the effect of different treatment strategies on mitochondrial function and to correlate in-vitro results to findings from in-vivo measurements of mitochondrial function. The authors hypothesize that interventional revascularization and therefore the restoration of blood and oxygen supply is more relevant to mitochondrial function compared to the effect of exercise training.

Patients with isolated pathologies of the superficial femoral artery and symptomatic PAD (Fontaine stage IIB) will be included and randomized to different treatment groups (conservative treatment versus interventional revascularization). Near-infrared refracted spectroscopy and the TIVITA ® hyperspectral camera will be used for in-vivo measurement of peripheral oxygen saturation and distal perfusion before and after an exercise. Muscle biopsies will be obtained from affected (gastrocnemius muscle) as well as from unaffected muscle (lateral vastus muscle) shortly before and 12 weeks after initiating treatment. Muscle samples will be investigated by measurement of CSA regarding mitochondrial content and HRR regarding mitochondrial respiration as well as for oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* Isolated flow limiting arteriosclerotic lesion of the superficial femoral artery
* Unilateral grade II b (Fontaine) peripheral arterial disease
* Informed consent

Exclusion Criteria:

* Flow limiting arteriosclerotic lesions of the infrarenal aorta, iliac arteries or common/ deep femoral artery
* Contraindication for exercise therapy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in mitochondrial function after defined treatment | After 12 weeks - compared to baseline at inclusion
  High-resolution respirometry of muscle biopsy sample
Change of near infrared spectroscopy | After 12 weeks - compared to baseline at inclusion
  Near infrared spectroscopy measurement of calf

SECONDARY OUTCOMES:
Change in flow mediated dilation of the brachial artery | After 12 weeks - compared to baseline at inclusion
  Evaluation of endothelial dysfunction with ultrasound measurements of flow mediated dilation of the brachial artery.
Change in standardized 6-minutes walking test | After 12 weeks - compared to baseline at inclusion
  Evaluation of cardiovascular risk with measurement of maximal walking distance (meters) in 6 minutes.
Change in ankle-brachial index | After 12 weeks - compared to baseline at inclusion
  Evaluation of hemodynamic parameters (ankle-brachial index).

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Wipper, MD, Study Chair — Medical University of Innsbruck
Locations (1):
- Medical University Innsbruck, Innsbruck, Tyrol, Austria

REFERENCES:
- [Derived] Schoenherr L, Heidler J, Kluckner M, Lobenwein D, Pesta D, Frese JP, Wipper SH, Gratl A. A Randomized Control Trial Investigating the Effect of Different Treatment Strategies on Mitochondrial Function in Peripheral Arterial Disease: A Study Protocol. J Surg Res. 2025 Mar;307:78-85. doi: 10.1016/j.jss.2025.01.014. Epub 2025 Feb 22. PMID 39987612